CLINICAL TRIAL: NCT03305575
Title: A Randomized Controlled Clinical Trial of Intrathecal Chloroprocaine vs. Bupivacaine for Cervical Cerclage
Brief Title: Intrathecal Chloroprocaine vs. Bupivacaine for Cervical Cerclage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12619
Record Dates: First submitted 2017-10-04; First posted 2017-10-10 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cervical Incompetence
Keywords: Cervical Cerclage; Bupivacaine; Chloroprocaine; spinal anesthesia
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesia provider responsible for the clinical care of the patient will be given an envelope prepared during randomization and instructed to open it and prepare the medication in a separate room, such that the investigator and patient cannot see which vial is being used to prepare the medication. The anesthesia provider will also be instructed not to reveal the allocation group to the investigator or the patient.
  Both bupivacaine and chloroprocaine are clear liquids, and the intended doses of both medications are the same volume, to insure complete blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chloroprocaine (Experimental): Patients assigned to chlorprocaine will receive a single spinal injection of 40 mg of chloroprocaine PF. (other name: pure Nesacaine MPF 3% in a total volume of 2ml)
  Interventions: Drug: Chloroprocaine
- Bupivacaine (Active Comparator): Patients assigned to bupivacaine will receive a single spinal injection of 7.5 mg of bupivacaine. (other name: pure Sensorcaine 0.75% diluted with normal saline to a total volume of 2ml).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Chloroprocaine — The patient will be randomly selected to receive either Chloroprocaine or Bupivacaine as the local medication for in spinal anesthesia, with a 50% chance to receive either drug.
  During the cervical cerclage procedure and in the recovery room, the patient will be checked for motor block (the ability to move feet and legs) and for sensory block(the ability to feel) using a plastic tip, every 5 minutes in the first hour, and at 10 minutes intervals afterwards until the anesthesia wears off completely. The patient will also be asked to walk and urinate after the local anesthetic wears off to ensure complete resolution of local anesthesia.
  Other Names: Sensorcaine
  Arms: Chloroprocaine
Drug: Bupivacaine — The patient will be randomly selected to receive either Chloroprocaine or Bupivacaine as the local medication for in spinal anesthesia, with a 50% chance to receive either drug.
  During the cervical cerclage procedure and in the recovery room, the patient will be checked for motor block (the ability to move feet and legs) and for sensory block(the ability to feel) using a plastic tip, every 5 minutes in the first hour, and at 10 minutes intervals afterwards until the anesthesia wears off completely. The patient will also be asked to walk and urinate after the local anesthetic wears off to ensure complete resolution of local anesthesia.
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
This study aims to compare the effect of chloroprocaine vs. bupivacaine on duration of motor block and duration until meeting discharge criteria in patients undergoing cervical cerclage. The hypothesis is that chloroprocaine will result in faster resolution of motor block.

DETAILED DESCRIPTION:
Cervical cerclage is an ambulatory surgical procedure of short duration commonly performed under spinal anesthesia. Bupivaciane and chlororpocaine are both commonly used, but how their use impacts clinical care, in particular patient flow, is not well studied.

This is a prospective, randomized, double blind, controlled trial. Participants meeting inclusion criteria will be randomly allocated to receive spinal anesthesia with either chloroprocaine or bupivacaine.

Patients will then be assessed for motor block and sensory level until they are discharged from the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification II or III females
* Age: 18-45 years old
* BMI ≤ 50 kg/m2
* Singleton pregnancy
* Simple prophylactic cervical cerclage
* Planning neuraxial anesthesia

Exclusion Criteria:

* Abdominal and complex cervical cerclage (e.g. bulging bag)
* Contraindication to neuraxial anesthesia
* Known hypersensitivity to chloroprocaine (a.k.a. Ester allergy), paraaminobenzoic acid (PABA) or bupivacaine (a.k.a. Amide allergy)
* Pseudocholinesterase deficiency
* Concomitant use with ergot-type oxytocic drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Drzymalski, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Concepcion M, Covino BG. Rational use of local anaesthetics. Drugs. 1984 Mar;27(3):256-70. doi: 10.2165/00003495-198427030-00005. PMID 6705717
- [Background] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878
- [Background] Yoos JR, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with small-dose bupivacaine in volunteers. Anesth Analg. 2005 Feb;100(2):566-572. doi: 10.1213/01.ANE.0000143356.17013.A1. PMID 15673895
- [Background] Casati A, Fanelli G, Danelli G, Berti M, Ghisi D, Brivio M, Putzu M, Barbagallo A. Spinal anesthesia with lidocaine or preservative-free 2-chlorprocaine for outpatient knee arthroscopy: a prospective, randomized, double-blind comparison. Anesth Analg. 2007 Apr;104(4):959-64. doi: 10.1213/01.ane.0000258766.73612.d8. PMID 17377114
- [Background] Beilin Y, Zahn J, Abramovitz S, Bernstein HH, Hossain S, Bodian C. Subarachnoid small-dose bupivacaine versus lidocaine for cervical cerclage. Anesth Analg. 2003 Jul;97(1):56-61, table of contents. doi: 10.1213/01.ane.0000068940.36040.54. PMID 12818944

RESULTS

PARTICIPANT FLOW:
Groups:
- Chloroprocaine: Patients assigned to chlorprocaine received a single spinal injection of 40 mg of chloroprocaine PF. (other name: pure Nesacaine MPF 3% in a total volume of 2ml)
- Bupivacaine: Patients assigned to bupivacaine received a single spinal injection of 7.5 mg of bupivacaine. (other name: pure Sensorcaine 0.75% diluted with normal saline to a total volume of 2ml).
Period: Overall Study
Arm/Group | Chloroprocaine | Bupivacaine
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chloroprocaine: Patients assigned to chlorprocaine will receive a single spinal injection of 40 mg of chloroprocaine PF. (other name: pure Nesacaine MPF 3% in a total volume of 2ml)
  Chloroprocaine: The patient will be randomly selected to receive either Chloroprocaine or Bupivacaine as the local medication for in spinal anesthesia, with a 50% chance to receive either drug.
  During the cervical cerclage procedure and in the recovery room, the patient will be checked for motor block (the ability to move feet and legs) and for sensory block(the ability to feel) using a plastic tip, every 5 minutes in the first hour, and at 10 minutes intervals afterwards until the anesthesia wears off completely. The patient will also be asked to walk and urinate after the local anesthetic wears off to ensure complete resolution of local anesthesia.
- Bupivacaine: Patients assigned to bupivacaine will receive a single spinal injection of 7.5 mg of bupivacaine. (other name: pure Sensorcaine 0.75% diluted with normal saline to a total volume of 2ml).
  Bupivacaine: The patient will be randomly selected to receive either Chloroprocaine or Bupivacaine as the local medication for in spinal anesthesia, with a 50% chance to receive either drug.
  During the cervical cerclage procedure and in the recovery room, the patient will be checked for motor block (the ability to move feet and legs) and for sensory block(the ability to feel) using a plastic tip, every 5 minutes in the first hour, and at 10 minutes intervals afterwards until the anesthesia wears off completely. The patient will also be asked to walk and urinate after the local anesthetic wears off to ensure complete resolution of local anesthesia.
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Bupivacaine | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4.5) | 29 (3.8) | 31 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 30.4 (5.9) | 29.7 (5.9) | 30 (5.4)
ASA [Mean (Standard Deviation); unit: Scores on a scale] — ASA classification ranges from I to V per the American Society of Anesthesiologists (ASA) as follow:
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation
  Scores on a scale | 2.3 (0.58) | 2 (0) | 2.1 (0.38)
Gestational age [Mean (Standard Deviation); unit: weeks] | 16 (3.9) | 14.8 (3.7) | 15.4 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Motor Block
Description: The time difference between local anesthetic injection and complete resolution of motor block -as measured on the Bromage scale:
  I = free movement of feet, legs and hip = No block II = able to flex knees, with free movement of feet = Mild block III = unable to flex knees, but with free movement of feet = Moderate block IV = unable to move legs or feet = Complete block
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Bupivacaine
Number analyzed (Participants) | 4 | 5
minutes | 75 (5.7) | 99 (48.0)

2. Secondary Outcome: Duration of Sensory Block
Description: The time difference between local anesthetic injection and complete resolution of sensory block. The sensory level was tested using a blunt needle tip along the patient's demratomal distribution of the spinal anesthetic.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Bupivacaine
Number analyzed (Participants) | 4 | 5
minutes | 127 (20.6) | 210 (56.1)

3. Secondary Outcome: Time to Ambulation
Description: The time difference between local anesthetic injection and patient's walking for the first time postoperatively.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Bupivacaine
Number analyzed (Participants) | 4 | 5
minutes | 110 (1.4) | 179 (2.6)

4. Secondary Outcome: Time to Micturation
Description: The time difference between local anesthetic injection and the patient's voiding for the first time postoperatively.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Bupivacaine
Number analyzed (Participants) | 4 | 5
minutes | 111 (1.3) | 233 (1.7)

ADVERSE EVENTS:
Time Frame: until the subjects were discharged form the post anesthesia care unit up to 6 hours.
Description: There were no adverse evens noted.
Arm/Group | Chloroprocaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03305575/Prot_SAP_000.pdf